CLINICAL TRIAL: NCT04263987
Title: A Comparison of Traditional and MOSES Laser Enucleation of the Prostate (MOLEP): A Prospective, Randomized, Double-blinded Control Trial
Brief Title: A Comparison of Traditional and MOSES Laser Enucleation of the Prostate (MOLEP): A Prospective, Randomized, Double-blinded Control Trial A Comparison of Traditional and MOSES Laser Enucleation of the Prostate (MOLEP): A Prospective, Randomized, Double-blinded Control Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Nicholas Kavoussi, Clinical Instructor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MOLEP Study
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Results first posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Holmium Laser Enucleation of Prostate (Active Comparator): Traditional holmium laser enucleation of the prostate as currently performed
  Interventions: Procedure: Moses laser enucleation of prostate
- Moses Holmium Laser Enucleation of Prostate (Experimental): holmium laser enucleation of the prostate as currently performed but with Moses laser settings activated.
  Interventions: Procedure: Moses laser enucleation of prostate

INTERVENTIONS:
Procedure: Moses laser enucleation of prostate — Using the moses settings with the Lumenis laser system to evaluate outcomes for enucleation of the prostate; hypothesis is that it leads to faster operative time

SUMMARY:
Holmium laser enucleation of the prostate (HOLEP) has proven to be efficacious and safe for the treatment of benign prostatic hypertrophy (BPH). New laser technologies such as the Moses Pulse laser system provide for improved energy delivery which may decrease blood loss and operative time. We seek to evaluate Moses technology for enucleation of the prostate in the setting of BPH.

DETAILED DESCRIPTION:
This is a single-center, prospective, double-blinded, randomized controlled trial comparing MOLEP to HOLEP. Inclusion criteria included all symptomatic BPH patients desiring enucleation with prostate sizes > 80ccs based on cross-sectional imaging. Patients are randomized in a 1:1 fashion and the study is powered to evaluate for a difference in operative time (i.e. alpha=0.05,N=21 per group). All surgeries will be performed with a 550 μm fiber. At the start of each case, a laser technician would be notified of randomization via envelope and randomize the settings to either Moses or traditional mode. The surgeons and patients were blinded to which mode was used. All surgeries will be performed using a two lobe technique and laser settings between 2J and 20-40Hz. Further recorded endpoints include change in blood loss, reduction in International Prostate Symptom Score (IPSS), improvement in uroflow parameters, and complications postoperatively at 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Any man with clinical symptoms fo BPH requiring surgery who has a prostate sized at greater than 80 grams

Exclusion Criteria:

* Anyone actively on anticoagulation perioperatively

Ages: 50 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — For prostatic disease
Enrollment: 60 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: VUMC 2019-2020
Period: Overall Study
Arm/Group | Holmium Laser Enucleation of Prostate | Moses Holmium Laser Enucleation of Prostate
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: men with benign prostatic hypertrophy (BPH)
Groups:
- Total: Total of all reporting groups
Arm/Group | Holmium Laser Enucleation of Prostate | Moses Holmium Laser Enucleation of Prostate | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (8) | 68 (6) | 69 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 30 | 30 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 25 | 25 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Operative Time
Description: time for surgery to take place
Time Frame: intraoperatively
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Holmium Laser Enucleation of Prostate | Moses Holmium Laser Enucleation of Prostate
Number analyzed (Participants) | 30 | 30
minutes | 101 (30) | 126 (22)

2. Secondary Outcome: Percentage of Change of Hematocrit
Description: Blood loss is calculated by the percentage of change of hematocrit
Time Frame: Baseline to postoperatively day 1
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Holmium Laser Enucleation of Prostate | Moses Holmium Laser Enucleation of Prostate
Number analyzed (Participants) | 30 | 30
percentage | 6 (4) | 9 (4)

ADVERSE EVENTS:
Time Frame: Up to 6 weeks postoperatively
Description: Adverse event information was collected for any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Holmium Laser Enucleation of Prostate | Moses Holmium Laser Enucleation of Prostate
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 4/30 | 3/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Holmium Laser Enucleation of Prostate (N=30) | Moses Holmium Laser Enucleation of Prostate (N=30)
cystitis (Renal and urinary disorders) | 4 (4) | 3 (3) — cystitis postoperatively, resolved with antibiotics

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-04-04): https://cdn.clinicaltrials.gov/large-docs/87/NCT04263987/Prot_001.pdf
  • Statistical Analysis Plan (2021-12-21): https://cdn.clinicaltrials.gov/large-docs/87/NCT04263987/SAP_002.pdf